CLINICAL TRIAL: NCT01188967
Title: A Double-Blind, Placebo-Controlled, Parallel Group Design Trial of the Selective D3 Antagonist, GSK598809, Added to CBT and NRT for Smoking Cessation and Prevention of Very Early Relapse to Smoking
Brief Title: Effectiveness of GSK598809, a Selective D3 Antagonist, Added to CBT and NRT for Smoking Cessation and Relapse Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Mclean Hospital (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Maurizio Fava, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIDA-19378-5; U01DA019378 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-26 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Nicotine Dependence
Keywords: Drugs, Investigational; Nicotine Dependence; Therapies for Relapse to Nicotine; Relapse Prevention; Smoking Cessation; Nicotine Cessation Therapies
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — GSK598809

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GSK598809 (Experimental): Active medication
  Interventions: Drug: GSK598809
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK598809 — Oral dose of 60 mg/day for a treatment period six weeks
  Arms: GSK598809
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to find out if an investigational drug, GSK598809 can help people who have very recently quit smoking; the investigators want to find out if continuing to take GSK598809 over six weeks can help prevent smokers from relapsing. To relapse means you "fall back" into smoking again after quitting. The investigators also want to find out if GSK598809 is safe to take without causing too many side effects.

DETAILED DESCRIPTION:
We propose to conduct a first test of the effect of the dopamine D3 receptor antagonist, GSK598809, on smoking behavior when treatment is started immediately following the quit date. To do this, we propose to conduct a 10-week, double-blind, placebo-controlled, proof of mechanism study in 90 adult smokers. Participants will complete baseline evaluations. They will receive manualized cognitive behavioral therapy, beginning prior to the quit date, and will set a quit date for the day before their week 2 study visit. They will be given short acting NRT (gum or lozenge) to use on their quit date. They will be asked to arrive for the week 2 visit with 18-24 hours abstinence and an expired air CO ≤ 10ppm. Those who do so will be randomly assigned to receive double blind GSK598809 or identical placebo for six weeks. Participants will begin double blind GSK598809 or placebo, both in conjunction with prn NRT up to 8 mg per day for two weeks. Participants will then continue double blind GSK598809 or placebo in the absence of NRT for 4 more weeks. At the end of this period (week 8 of the study), participants will then be followed 2 weeks after discontinuation of double blind treatment to complete the 10 weeks of the study.

ELIGIBILITY:
Exclusion criteria:

1. Pregnant or able to become pregnant and not willing to use approved contraception.
2. Breastfeeding or planning to breastfeed during the study or lactating within the month prior to enrollment.
3. Has any of the following medical conditions/situations:

   Severe or unstable COPD or Asthma Bundle branch block Evidence of active neurological disease, including current migraine headaches requiring chronic treatment.

   Clinically significant renal dysfunction eGFR <60 History of any tissue/organ transplant Total fasting cholesterol or triglycerides greater than 2 times the upper limit of normal Previous or current history of cancer, including skin cancer Serum Prolactin > 25 ng/mL at the time of screening or randomization Evidence of chronic liver disease or ALT, AST, or alkaline phosphatase values >1.5 times the upper limit of normal, total bilirubin values > the upper limit of normal, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C) Positive screening Hepatitis B surface antigen or Hepatitis C antibody, or positive result within 3 months of screening A positive test for HIV antibody Any other unstable cardiovascular or pulmonary disease, or medication for said diseases has been changed in the past 3 months, or the medication is listed on the excluded medications list.
4. Is unlikely to cooperate or unable to follow all of the procedures outlined in the protocol
5. Use of tobacco-containing products other than cigarettes (e.g., cigar, pipe) and unwilling to discontinue use of these on the quit date.
6. Abuse or dependence of any substance other than nicotine or caffeine in the past 6 months.
7. Diagnosis of major depressive disorder in the past 6 months.
8. Lifetime DSM-IV diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, bipolar disorder, delusional disorder or psychotic disorders not elsewhere classified as determined by SCID.
9. History of multiple adverse drug reactions.
10. Has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
11. Urine positive for drugs of abuse at screening and any pre-randomization visit.
12. Alcohol abuse, defined as self-report of an average weekly intake of > 21 standard drinks or an average daily intake of >3 standard drinks (males) or an average weekly intake of >14 standard drinks or an average daily intake of >2 standard drinks (females) in the past 6 months. One unit is equivalent to a half-pint (220mL) of beer or one (25mL) measure of spirits or one glass (125mL) of wine. Participants will be advised to minimize alcohol consumption during the study, as there may be the potential for additive effects of study medication and alcohol, potentially causing greater sedation and feeling of intoxication than alcohol alone.
13. Has been exposed to more than four new chemical entities within 12 months prior to the first day of the double-blind treatment phase.
14. Has used non-prescription drugs or herbal medicines that are centrally active within 14 days prior to the first dosing day, with the exception of non-daily PRN use of acetaminophen or ibuprofen and daily use of vitamins.
15. Has ever used chronic antipsychotic, anti-epileptic, or mood stabilizing medication; has used anti-anxiety medication, antidepressant medication, or prescription sedatives or hypnotics within 5 half lives or two weeks of randomization, whichever is greater.
16. Has a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator makes participation contraindicated.
17. Has donated blood such that participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56-day period.
18. Has a failed smoking cessation attempt using adequate smoking cessation pharmacotherapy within the last month.
19. Current Axis II DSM-IV diagnosis that may interfere with the conduct of the study.
20. Personal or family history of long QT syndrome, personal or family history of unexplained syncope, or family history of unexplained sudden death.
21. Currently using, or have used within the month prior to study start, any drug that can cause prolongation of the QT interval.
22. Currently using any HMG CoA Reductase Inhibitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital; Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 84 participants signed consent and 40 of those participants were found ineligible. 11 participants voluntarily withdrew consent. 4 participants were terminated by the investigator for reasons other than toxicity/adverse events (ie noncompliance). 11 participants were lost to follow up.
Groups:
- GSK598809 Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects will be randomized with a block size of 4. This group received 60 mg GSK598809 pills, the active treatment, for 6 weeks.
- Placebo Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects will be randomized with a block size of 4. This group received placebo pills.
Period: Overall Study
Arm/Group | GSK598809 Treatment Group | Placebo Group
Started | 10 | 8
Completed | 5 | 4
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects were randomized with a block size of 4. This group received placebo pills.
- GSK598809 Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects were randomized with a block size of 4. This group received the active treatment: GSK598809 pills,60 mg/day.
- Total: Total of all reporting groups
Arm/Group | Placebo Treatment Group | GSK598809 Treatment Group | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants] — The study only included participants aged 18-65.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 8 | 10 | 18
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — The study only included participants aged 18-65
  years | 48.7 (5) | 46.7 (5) | 47.7 (5)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: 4-week, Continuous Tobacco Abstinence at the End of the 6-week, Double Blind, Treatment Phase
Description: The hypothesis is that those assigned to GSK598809 will demonstrate a higher rate of biochemically-verified, 4-week, continuous tobacco abstinence than those assigned to identical placebo at the end of the 6-week, double blind, treatment phase. Four-week continuous abstinence will be defined as Timeline Followback Calendar confirmation at study visit of smoking no cigarettes in the past 7 days, and expired air CO<10ppm for 4 consecutive weeks (the last 4 weeks of the randomized phase)
Time Frame: Week 8 of the study
Population: 9 participants completed this visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Treatment Group | GSK598809 Treatment Group
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

2. Secondary Outcome: 7-day, Point-prevalence Tobacco Abstinence at the End of the First Week of Exposure to GSK598809/Placebo
Description: The hypothesis is that those assigned to GSK598809 will demonstrate a higher rate of biochemically-verified, 7-day, point-prevalence tobacco abstinence than those assigned to identical placebo at the end of the first week of exposure to GSK598809/placebo.
Time Frame: Week 3 of the study
Population: 13 participants completed week 1 visit
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects will be randomized with a block size of 4. This group received placebo pills.
- GSK598809 Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects will be randomized with a block size of 4. This group received GSK598809 pills, the active treatment.
Arm/Group | Placebo Treatment Group | GSK598809 Treatment Group
Number analyzed (Participants) | 6 | 7
Participants | 2 | 0

3. Secondary Outcome: 7-day, Point-prevalence Tobacco Abstinence at the End of 6 Weeks Exposure to GSK598809/Placebo
Description: The hypothesis is that those assigned to GSK598809 will demonstrate a higher rate of biochemically-verified, 7-day, point-prevalence tobacco abstinence than those assigned to identical placebo at the end of 6 weeks exposure to GSK598809/placebo.
Time Frame: Week 8 of the study
Population: 7 participants completed week 6 weeks exposure to GSK598809/placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Treatment Group | GSK598809 Treatment Group
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With 7-day, Point-prevalence Tobacco Abstinence 2-weeks After Discontinuation of Double Blind Study Medications
Description: The hypothesis is that those assigned to GSK598809 will demonstrate a higher rate of biochemically-verified, 7-day, point-prevalence tobacco abstinence than those assigned to identical placebo two weeks after discontinuation of double blind study medications.
  7-day, Point-prevalence tobacco abstinence was defined as not smoking for the 7 consecutive days before this visit after discontinuation of double blind study medications
Time Frame: Week 10 of the study
Population: 7 participants completed this visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Treatment Group | GSK598809 Treatment Group
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study, 10 weeks in total (2 weeks before quitting, 6 weeks on double blind GSK598809 or placebo, 2 weeks of follow up).
Description: Adverse events were recorded for all subjects at weekly sessions.
Groups:
- Placebo Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects will be randomized with a block size of 4. This group received the placebo pills.
- GSK598809 Treatment Group: There is a 6-week, double-blind, placebo-controlled randomized treatment phase to evaluate the effect of study medication on craving, abstinence, and lapses to smoking. Eligible subjects will be randomized with a block size of 4. This group received the GSK598809 pills, the active treatment.
Arm/Group | Placebo Treatment Group | GSK598809 Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/10
Other Adverse Events (participants affected / at risk) | 4/8 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Group (N=8) | GSK598809 Treatment Group (N=10)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) — The subject notified the clinic on 8/25/11 that he was unable to attend his weekly visit because he was hospitalized for an anal abscess.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Group (N=8) | GSK598809 Treatment Group (N=10)
Leg Cramps (General disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (1) | 0 (0)
Fungal Skin Infection (General disorders) | 0 (0) | 1 (1)
Urinary Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 2 (2) | 1 (1)
Peripheral Vascular Disease (General disorders) | 0 (0) | 1 (1)
Weight Gain (General disorders) | 1 (1) | 0 (0)
Dry Tongue (General disorders) | 0 (0) | 1 (1)
Numbness of Tongue (General disorders) | 0 (0) | 1 (1)
Chest Tightness (General disorders) | 0 (0) | 1 (1)
Eczema Flame (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
URI (Renal and urinary disorders) | 2 (2) | 1 (1)
Cold (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less